CLINICAL TRIAL: NCT02973139
Title: Fibrinolytic Therapy Versus Medical Thoracoscopy for Treatment of Pleural Infection: A Randomized Clinical Trial
Brief Title: Fibrinolysis Compared to Thoracoscopy for Pleural Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Adnan Majid, MD FCCP, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000307
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Pleural Infection; Pleural Diseases
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracoscopy group (Active Comparator): Patients randomized to the Thoracoscopy group will undergo medical thoracoscopy.
  Interventions: Other: Medical Thoracoscopy
- Fibrinolytic group (Active Comparator): Patients randomized to the Fibrinolytic group will receive intrapleural therapy of combined tissue plasminogen activator (tPA) and human recombinant deoxyribonuclease (DNase)
  Interventions: Other: Fibrinolytic Group

INTERVENTIONS:
Other: Medical Thoracoscopy — Medical thoracoscopy will be performed as per standard protocols.
  Arms: Thoracoscopy group
Other: Fibrinolytic Group — Patients will receive intrapleural combination of TPA (10 mg) and DNAse (5 mg). Therapy will be given twice daily for a maximum of 6 doses
  Arms: Fibrinolytic group

SUMMARY:
The purpose of this prospective randomized clinical trial is to compare two currently accepted standard-of-care treatment strategies: Medical thoracoscopy as compared to instillation of intrapleural tissue Plasminogen Activator (TPA) and human recombinant Deoxyribonuclease (DNase) for the management of empyema or complex parapneumonic effusion (CPPE) in adults.

DETAILED DESCRIPTION:
Background: Pleural infection (empyema or complex parapneumonic effusion (CPPE)) represents one of the most common clinical diagnoses encountered in clinical practice in the United States (US) It is associated with substantial morbidity and mortality despite advances in medical diagnostic and therapeutic strategies.

Objective: Compare two standard of care treatments: TPA/DNase vs early medical Thoracoscopy

Methods: We will conduct a prospective randomized clinical trial. We plan to enroll a total of 80 patients and randomize them to either Medical Thoracoscopy group or Fibrinolytic Therapy group.

Follow-up will be daily until hospital discharge and at 6 and 12 weeks in the outpatient setting

Primary Outcome: Duration of hospital stay after intervention

Secondary Outcome: Failure rate of assigned treatment and adverse events

Potential Outcome and Benefit: Determine best strategy for treating patients with pleural infection

ELIGIBILITY:
Inclusion Criteria:

* Subjects >18 years old with:
* Evidence of empyema or complex parapneumonic effusion

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Inability to give informed written consent
* Previous thoracic surgery or thrombolytic therapy for pleural infection
* Medical thoracoscopy cannot be performed within 48 hours
* Hemodynamic instability or severe hypoxemia
* Non corrected coagulopathy
* Homogeneously echogenic effusion on pleural ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay after intervention | 12 week follow up period
  Number of days hospitalized

SECONDARY OUTCOMES:
Number of days with chest drainage | 12 week follow up period
  Number of days with chest drainage
Total length of hospital stay | 12 week follow up period
  Total days spent in the hospital
Failure rate of assigned treatment necessitating intervention | 12 week follow up period
  defined as any of the following:
  1. Surgical intervention (VATS, open thoracotomy) in the medical thoracoscopy or fibrinolytic therapy arm
  2. Need of additional chest tube and/or fibrinolytic therapy in the medical thoracoscopy arm due to clinical non-responsiveness
  3. Need of additional chest tube in the fibrinolytic therapy arm due to clinical non-responsiveness
Adverse events | 12 week follow up period
  Any adverse event (pain or bleeding)
In hospital and 30-day mortality | 30 days
  Death of a patient while being hospitalized or up to 30 days after
Change in pleural fluid volume on Chest CT scan prior to randomization (day 0) to prior to chest tube removal measured by radiologist blinded to treatment allocation using image J software | 12 week follow up period
  Pleural fluid volume measured with CT scan
Inflammatory biomarker (CRP) from randomization (day 0), at 6 weeks and 12 weeks respectively | at randomization and at 6 and12 week follow up visit
  Inflammatory biomarker measure
Total costs of each treatment modality | 6 and 12 week follow up period
  Total cost of each of treatment modality

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kheir F, Thakore S, Mehta H, Jantz M, Parikh M, Chee A, Kaphle U, Sisnega C, Fernandez-Bussy S, Majid A. Intrapleural Fibrinolytic Therapy versus Early Medical Thoracoscopy for Treatment of Pleural Infection. Randomized Controlled Clinical Trial. Ann Am Thorac Soc. 2020 Aug;17(8):958-964. doi: 10.1513/AnnalsATS.202001-076OC. PMID 32421353